CLINICAL TRIAL: NCT07248059
Title: Prevalence of Oral Findings in Egyptian Patients Diagnosed With Familial Mediterranean Fever: A Hospital-Based Cross-sectional Study
Brief Title: Prevalence of Oral Findings in Egyptian Patients Diagnosed With Familial Mediterranean Fever
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amr Mahmoud Almorsy Ahmed, MSc candidate at the Oral Medicine and Periodontology department, Faculty of dentistry, Cairo university, Cairo University
Other Study IDs: OMED 2-1-1
Record Dates: First submitted 2025-09-23; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-09

CONDITIONS: Familial Mediterranean Fever (FMF ) and Oral Findings
Keywords: FMF , Oral lesions
MeSH Terms: conditions — Familial Mediterranean Fever

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Egyptian children with FMF: Egyptian children aged 6 to 15 years, with a confirmed diagnosis of Familial Mediterranean Fever (FMF), attending the Collagen Diseases Clinic at Abu Elreesh Japanese Children's Hospital.

SUMMARY:
This is an observational descriptive cross-sectional study will be performed at the Collagen Diseases Clinic, Abu Elreesh Japanese Children's Hospital, Cairo, Egypt. This study aims to Investigate and assess the prevalence of oral findings or lesions in Egyptian patients diagnosed with FMF

DETAILED DESCRIPTION:
Familial Mediterranean Fever (FMF) is a monogenic autoinflammatory disease and the most common of the periodic fever syndromes. FMF patients usually present with recurrent episodes of fever. They also suffer from abdominal, chest and joint pain due to serositis. Patients may present with erysipelas, amyloidosis, and rarely, ophthalmic manifestations. The oral cavity and related facial structures may also be affected. Oral lesions such as: recurrent oral ulcers, macroglossia and high arched palate. The prevalence of oral findings in FMF remains variable and underexplored. An accurate examination is required for the early identification of FMF cases. Diagnostic delay is common in FMF and complicated by incomplete clinical presentation and overlap in symptoms with other diseases. So, Recognizing other signs and symptoms could be incorporated into diagnostic criteria of FMF for early diagnosis and treatment with improvement of quality of life. This study will be performed at the Collagen Diseases Clinic, Abu Elreesh Japanese Children's Hospital, Cairo, Egypt. Egyptian children aged 6 to 15 years, with a confirmed diagnosis of FMF will be enrolled and recruited consecutively either at their initial diagnosis or follow-up visits. On the other hand, Children with other systemic diseases not related to FMF, children who are unable to cooperate or refuse to participate will be excluded from the study. During this visit, data will be collected through clinical oral examination using a standardized dental chart, along with a review of their medical records. The oral findings will be reported as binary data (yes / no). Moreover, documenting such oral findings could provide an important baseline for identifying FMF-associated anomalies in the population.

ELIGIBILITY:
Inclusion Criteria:

* Egyptian children aged 6 to 15 years
* Children with a confirmed diagnosis of Familial Mediterranean Fever (FMF)
* Children attending the Collagen Diseases Clinic at Abu Elreesh Japanese Children's Hospital.

Exclusion Criteria:

* Children with other systemic diseases not related to FMF
* Children who are unable to cooperate or refuse to participate

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Egyptian children aged 6 to 15 years, with a confirmed diagnosis of Familial Mediterranean Fever (FMF), attending the Collagen Diseases Clinic at Abu Elreesh Japanese Children's Hospital will be enrolled and recruited consecutively at a one point in time.
Sampling Method: Non-Probability Sample
Enrollment: 359 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-10-30 (Estimated); Study Completion 2027-07-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Oral Findings in Egyptian patients Diagnosed with Familial Mediterranean Fever | At enrollment ( single cross-sectional visit)
  The data will be collected through clinical oral examination using a standardized dental chart, along with a review of their medical records. The oral findings including high-arched palate, enamel defects, macroglossia, recurrent oral ulcers, and short philtrum will be reported as binary data (yes / no). Binary data such as prevalence of oral manifestations will be reported as a proportion.

CONTACTS AND LOCATIONS:
Overall Officials: Fat'heya Mohamed Zahran, Professor, Principal Investigator — Cairo University; noha adel ibrahim, lecturer, Study Chair — Cairo University; Hend mohamed abu shaday, assistant professor, Study Chair — Cairo University
Locations (1):
- Collagen Diseases Clinic, Abu Elreesh Japanese Children's Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No